CLINICAL TRIAL: NCT02642029
Title: Cerebellar Transcranial Magnetic Stimulation (cTMS) in Psychotic Disorders: Effect on Time Perception, Executive Function, and Mood and Psychotic Symptoms
Brief Title: Targeting Cerebellum to Treat Psychosis: a Transcranial Magnetic Stimulation (TMS) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ann K Shinn, Assistant Professor, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015P001833
Record Dates: First submitted 2015-11-20; First posted 2015-12-30 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder I
Keywords: time perception; executive function; psychosis; mood symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intermittent TBS (iTBS) (Experimental): Single session of intermittent theta-burst stimulation (600 pulses in blocks of 2s, separated by 8s of pause) to cerebellar vermis.
  Interventions: Device: Excitatory TMS
- Continuous TBS (cTBS) (Active Comparator): Single session of continuous theta-burst stimulation of 600 pulses to cerebellar vermis.
  Interventions: Device: Inhibitory TMS
- Sham TBS (Sham Comparator): Single session, using the exact same procedures as the active arms but with a sham coil, which is designed to induce the same nonspecific sensory effects of TMS (auditory and somatosensory activation) without inducing the neuromodulatory magnetic fields.
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: Excitatory TMS — Single session of intermittent theta-burst stimulation (600 pulses in blocks of 2s, separated by 8s of pause) to cerebellar vermis.
  Other Names: iTBS
  Arms: Intermittent TBS (iTBS)
Device: Inhibitory TMS — Single session of continuous theta-burst stimulation of 600 pulses to cerebellar vermis.
  Other Names: cTBS
  Arms: Continuous TBS (cTBS)
Device: Sham TMS — Single session, using the exact same procedures as the active arms but with a sham coil, which is designed to induce the same nonspecific sensory effects of TMS (auditory and somatosensory activation) without inducing the neuromodulatory magnetic fields.
  Other Names: shamTBS
  Arms: Sham TBS

SUMMARY:
The goal of this study is to use transcranial magnetic stimulation (TMS) to investigate the impact of modulating cerebellar activity on time perception, executive function, and mood and psychotic symptoms in psychosis patients (i.e., schizophrenia, schizoaffective disorder, and bipolar disorder with psychotic features). The investigators hypothesize that abnormally reduced activity in the cerebellum contributes to the abnormalities in patients, that cerebellum-mediated disruptions in time perception may partially underlie executive dysfunction and symptoms, and that cerebellar stimulation will normalize disease-relevant outcome measures.

DETAILED DESCRIPTION:
The cerebellum plays a major role in integrative processing of higher order cognitive and affective functions, but it has not been considered a major treatment target for psychotic disorders. The goal of this study is to administer three different conditions of transcranial magnetic stimulation (TMS)-- excitatory, inhibitory, and sham TMS-- in a cross-over design in psychosis patients (i.e., schizophrenia, schizoaffective disorder, and bipolar disorder with psychotic features) to investigate with causal explanatory power the role of the cerebellum as a treatment target for psychotic disorders. More specifically, the investigators will measure the effects of cerebellar excitation and inhibition on time perception, executive function, and symptomatology. TMS will be administered using a theta-burst stimulation (TBS) protocol applied to the posterior cerebellar vermis. Participants will undergo three study sessions, one for each of the three TMS conditions. During each session, the investigators will administer validated cognitive paradigms and clinical measures immediately before and after TMS.

The specific aims are to:

1: Investigate the role of the cerebellum in abnormalities of time perception, executive function, and mood and psychotic symptoms by evaluating these functions before and immediately after excitatory, inhibitory, or sham TMS applied to the cerebellar vermis in patients with psychosis.

(1a) Time perception hypothesis: Patients with psychotic disorders will have impaired timing perception, i.e., higher number of errors and/or greater inter-trial variability in an interval discrimination task both at baseline and after sham TMS. The investigators predict that the abnormalities in patients will improve after excitatory but not inhibitory TMS.

(1b) Executive function hypothesis: Patients will show a higher number of errors and longer reaction times on the N-back working memory task, both at baseline and after sham TMS. The investigators predict that these deficits in patients will improve after excitatory but not inhibitory TMS.

(1c) Symptom hypothesis: Symptom ratings using visual analog scales will improve in the period immediately after excitatory but not inhibitory TMS, and show no significant change after sham TMS.

2: Investigate the relationship between time perception and symptomatology in patients with psychotic disorders. Hypothesis: The investigators predict that performance on the time perception task will correlate with performance on a working memory task as well as with mood and psychotic symptoms.

This study may improve understanding about the role of the cerebellum in the pathophysiology of psychotic disorders. Such knowledge can potentially guide the development of cerebellar TMS as a therapeutic intervention for psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  * Men and women
  * Ages 18-50 years
  * Patients diagnosed with schizophrenia (SZ), schizoaffective disorder (SZA), or psychotic bipolar disorder (BP).
  * On a stable psychiatric medication regimen for at least a month prior to and during study participation
* Healthy Controls:

  * Men and women
  * Ages 18-50 years
  * Without major psychiatric illness

Exclusion Criteria:

* Patients

  * Any change in psychiatric medications within a month prior to and during study participation
  * Legal or mental incompetency
  * Intellectual disability
  * Substance use disorder (abuse or dependence) with active use within the last 3 months
  * Significant medical or neurological illness
  * Prior neurosurgical procedure
  * History of seizures
  * History of electroconvulsive therapy (ECT) or clinical TMS within the past three months
  * History of participation in a cerebellar TMS study
  * Implanted cardiac pacemakers
  * Patients who have conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head or neck, or are non-removable and within 30 cm of the treatment coil. These include:

    * Aneurysm clips or coils
    * Carotid or cerebral stents
    * Metallic devices implanted in the head (e.g. Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculo-peritoneal shunt)
    * Magnetically active dental implants
    * Cochlear/otologic implants
    * CSF shunts
    * Ferromagnetic ocular implants
    * Pellets, bullets, fragments less than 30 cm from the coil
    * Facial tattoos with metallic ink, permanent makeup less than 30 cm from the coil
  * Pregnant women
* Healthy Controls:

  * History of major psychiatric illness, including psychosis
  * Has a first-degree relative with psychosis
  * Active use of psychotropic medications
  * Legal or mental incompetency
  * Intellectual disability
  * Substance use disorder (abuse or dependence) with active use within the last 3 months
  * Significant medical or neurological illness
  * Prior neurosurgical procedure
  * History of seizures
  * History of ECT treatment or clinical TMS within the past three months
  * History of participation in a cerebellar TMS study
  * Implanted cardiac pacemakers
  * Individuals who have conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head or neck, or are non-removable and within 30 cm of the treatment coil. These include:

    * Aneurysm clips or coils
    * Carotid or cerebral stents
    * Metallic devices implanted in the head (e.g. Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, transcutaneous electrical nerve stimulation (TENS) unit, or ventriculo-peritoneal shunt)
    * Magnetically active dental implants
    * Cochlear/otologic implants
    * Cerebrospinal fluid (CSF) shunts
    * Ferromagnetic ocular implants
    * Pellets, bullets, fragments less than 30 cm from the coil
    * Facial tattoos with metallic ink, permanent makeup less than 30 cm from the coil
  * Pregnant women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann K Shinn, MD, MPH, Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts

REFERENCES:
- [Derived] Shinn AK, Hurtado-Puerto AM, Roh YS, Ho V, Hwang M, Cohen BM, Ongur D, Camprodon JA. Cerebellar transcranial magnetic stimulation in psychotic disorders: intermittent, continuous, and sham theta-burst stimulation on time perception and symptom severity. Front Psychiatry. 2023 Nov 13;14:1218321. doi: 10.3389/fpsyt.2023.1218321. eCollection 2023. PMID 38025437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: N=28 participants were enrolled (provided informed consent to participate in the study).
  (Note: when I enter the number in the "Protocol Enrollment" field, the number does not save.)
Pre-assignment Details: Two participants did not undergo TBS after enrollment. N=1 participant enrolled and completed the pre-intervention clinical evaluation but withdrew prior to randomization (no specific reason given by the participant). N=1 participant had a positive urine drug screen after enrollment; as active substance use within the prior 3 months is an exclusion criterion, the participant was excluded prior to randomization.
Groups:
- Sham-iTBS-cTBS: Randomized first to Sham. Then randomized to iTBS for the second study visit. Then randomized to cTBS for the third study visit.
- Sham-cTBS-iTBS: Randomized first to Sham. Then randomized to cTBS for the second study visit. Then randomized to iTBS for the third study visit.
- iTBS-sham-cTBS: Randomized first to iTBS. Then randomized to sham for the second study visit. Then randomized to cTBS for the third study visit.
- iTBS-cTBS-sham: Randomized first to iTBS. Then randomized to cTBS for the second study visit. Then randomized to sham TBS for the third study visit.
- cTBS-sham-iTBS: Randomized first to cTBS. Then randomized to sham for the second study visit. Then randomized to iTBS for the third study visit.
- cTBS-iTBS-sham: Randomized first to cTBS. Then randomized to iTBS for the second study visit. Then randomized to sham TBS for the third study visit.
Period: Study Visit 1 (1 Day)
Arm/Group | Sham-iTBS-cTBS | Sham-cTBS-iTBS | iTBS-sham-cTBS | iTBS-cTBS-sham | cTBS-sham-iTBS | cTBS-iTBS-sham
Started | 6 (N=11 total participants were randomized to sham for the first study visit. For study visit 1, participants could be randomized to ONE OF THREE interventions (iTBS, cTBS, or sham TBS), not one of six interventions as this participant flow section suggests. The total number randomized to sham is the number started in "Sham-iTBS-cTBS" PLUS the number started in "Sham-cTBS-iTBS.") | 5 (N=11 total participants were randomized to sham for the first study visit. For study visit 1, participants could be randomized to ONE OF THREE interventions (iTBS, cTBS, or sham TBS), not one of six interventions as this participant flow section suggests. The total number randomized to sham is the number started in "Sham-iTBS-cTBS" PLUS the number started in "Sham-cTBS-iTBS.") | 3 (N=7 total participants were randomized to iTBS for the first study visit. For study visit 1, participants could be randomized to ONE OF THREE interventions (iTBS, cTBS, or sham TBS), not one of six interventions as this participant flow section suggests. The total number randomized to sham is the number started in "iTBS-sham-cTBS" PLUS the number started in "iTBS-cTBS-sham.") | 4 (N=7 total participants were randomized to iTBS for the first study visit. For study visit 1, participants could be randomized to ONE OF THREE interventions (iTBS, cTBS, or sham TBS), not one of six interventions as this participant flow section suggests. The total number randomized to sham is the number started in "iTBS-sham-cTBS" PLUS the number started in "iTBS-cTBS-sham.") | 4 (N=8 total participants were randomized to cTBS for the first study visit. For study visit 1, participants could be randomized to ONE OF THREE interventions (iTBS, cTBS, or sham TBS), not one of six interventions as this participant flow section suggests. The total number randomized to sham is the number started in "cTBS-sham-iTBS" PLUS the number started in "cTBS-iTBS-sham.") | 4 (N=8 total participants were randomized to cTBS for the first study visit. For study visit 1, participants could be randomized to ONE OF THREE interventions (iTBS, cTBS, or sham TBS), not one of six interventions as this participant flow section suggests. The total number randomized to sham is the number started in "cTBS-sham-iTBS" PLUS the number started in "cTBS-iTBS-sham.")
Completed | 6 | 5 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1 (≥ 36 Hours)
Arm/Group | Sham-iTBS-cTBS | Sham-cTBS-iTBS | iTBS-sham-cTBS | iTBS-cTBS-sham | cTBS-sham-iTBS | cTBS-iTBS-sham
Started | 6 | 5 | 3 | 4 | 4 | 4
Completed | 5 | 4 | 3 | 4 | 3 | 4
Not Completed | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol violation: Excluded due to change in psychiatric medications | 0 | 0 | 0 | 0 | 1 | 0
Period: Study Visit 2 (1 Day)
Arm/Group | Sham-iTBS-cTBS | Sham-cTBS-iTBS | iTBS-sham-cTBS | iTBS-cTBS-sham | cTBS-sham-iTBS | cTBS-iTBS-sham
Started | 5 (Of the 9 participants who completed sham TBS, 5 were randomized to iTBS for the second study visit.) | 4 (Of the 9 participants who completed sham TBS, 4 were randomized to cTBS for the second study visit.) | 3 (Of the 7 participants who completed iTBS, 3 were randomized to sham TBS for the second study visit.) | 4 (Of the 7 participants who completed iTBS, 4 were randomized to cTBS for the second study visit.) | 3 (Of the 7 participants who completed cTBS, 3 were randomized to sham TBS for the second study visit.) | 4 (Of the 7 participants who completed cTBS, 4 were randomized to iTBS for the second study visit.)
Completed | 4 | 4 | 3 | 4 | 3 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout 2 (≥ 36 Hours)
Arm/Group | Sham-iTBS-cTBS | Sham-cTBS-iTBS | iTBS-sham-cTBS | iTBS-cTBS-sham | cTBS-sham-iTBS | cTBS-iTBS-sham
Started | 4 | 4 | 3 | 4 | 3 | 4
Completed | 2 | 4 | 3 | 4 | 3 | 4
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Excluded due to hospitalization for substance misuse | 1 | 0 | 0 | 0 | 0 | 0
Period: Study Visit 3 (1 Day)
Arm/Group | Sham-iTBS-cTBS | Sham-cTBS-iTBS | iTBS-sham-cTBS | iTBS-cTBS-sham | cTBS-sham-iTBS | cTBS-iTBS-sham
Started | 2 | 4 | 3 | 4 | 3 | 4
Completed | 2 | 4 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- All Study Participants: All enrolled participants (study was designed for all participants to receive all 3 interventions- iTBS, cTBS, and sham TBS).
Arm/Group | All Study Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 1
  Unknown or Not Reported | 0
Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia | 6
  Schizoaffective disorder | 12
  Bipolar disorder with psychotic features | 10
Education [Count of Participants; unit: Participants]
  High School/GED | 6
  Part-college or 2-year college | 10
  College/bachelor's degree | 8
  Graduate/professional school | 4
Estimated Intelligence Quotient (IQ) [(North American Adult Reading Test (NAART)] [Mean (Standard Deviation); unit: units on a scale] — The North American Adult Reading Test (NAART) is a quickly administered index that is widely used to estimate verbal intellectual ability (Uttl, J Clin & Exper Neuropsychology 2002). It consists of 61 irregular rare words scored for accuracy according to North American pronunciation rules. The NAART has been used to estimate Weschler Adult Intelligence Scale, Revised (WAIS-R) verbal IQ, performance IQ, and full scale IQ (Blair & Spreen, Clinical Neuropsychologist 1989). Higher values represent higher intellectual ability. Population average IQ is 100; 68% of scores fall between 85 and 115.
  units on a scale
    Verbal IQ | 118.3 (10.4)
    Performance IQ | 114.5 (4.9)
    Full scale IQ | 118.7 (9.1)
Positive and Negative Syndrome Scale (PANSS) [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS; Kay et al., Schizoph. Bulletin 1987) is a widely used standardized measure to assess the severity of psychotic symptoms. The scale is interviewer-rated and consists of 30 items (7 positive, 7 negative, and 16 general psychopathology symptoms). Each item is rated on a scale from 1 ("absent") to 7 ("extreme"). Items in each of the sub-scales are summed to produce the positive (range 7-49), negative (range 7-49), and general psychopathology (range 16-112) subscores. The sum of all PANSS items yields the PANSS total score (range 30-210).
  units on a scale
    PANSS, total | 41.0 (27.3)
    PANSS, positive | 9.8 (7.3)
    PANSS, negative | 10.4 (7.3)
    PANSS, general psychopathology | 20.9 (13.5)
Young Mania Rating Scale (YMRS) [Mean (Standard Deviation); unit: units on a scale] — The Young Mania Rating Scale (YMRS; Young et al., Br J Psychiatry 1978) is a widely used standardized measure to assess the severity of manic symptoms. The scale is interviewer-rated and consists of 11 items. Seven items (elevated mood, increased motor activity/energy, sexual interest, sleep, thought disorder, appearance, insight) are rated on a Likert scale from 0 to 4. Four items (irritability, speech, content, disruptive/aggressive behavior) are rated from 0 to 8. Item scores are summed to produce the total score (range 0 to 60). Higher scores indicate greater severity of manic symptoms.
  units on a scale | 7.3 (9.3)
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS; Montgomery & Asberg, Br J Psychiatry 1979) is a widely used standardized measure to assess the severity of depressive symptoms. The MADRS is interviewer-rated and consists of 10 items. Each item is rated on a Likert scale from 0 to 6. Item scores are summed to produce the total score (range 0 to 60). Higher scores indicate greater severity of depressive symptoms.
  units on a scale | 10.9 (11.2)
Psychotic Symptom Rating Scale (PSYRATS-AH) [Mean (Standard Deviation); unit: units on a scale] — The auditory hallucination (AH) sub-scale of the Psychotic Symptom Rating Scale (PSYRATS; Haddock et al., Psychol Med 1999) is an interviewer-administered AH measure that is widely used in AH research. The PSYRATS-AH assesses 11 AH characteristics of AH (e.g., frequency, duration, loudness, degree of distress, controllability), with each item rated on a Likert scale from 0-4 (total range 0-44). Higher scores on the PSYRATS-AH indicate greater severity of auditory hallucinations.
  units on a scale | 4.1 (9.4)
Chlorpromazine equivalent dose (CPZ) [Mean (Standard Deviation); unit: mg/day] | 242.4 (311.6)
Taking antipsychotic medication [Count of Participants; unit: Participants] | 17
Taking mood stabilizer [Count of Participants; unit: Participants] | 14
Taking either antipsychotic or mood stabilizer [Count of Participants; unit: Participants] | 23
Not taking any psychotropic medication [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Change (Δ) in Accuracy of Time Interval Discrimination Pre- and Post-TMS
Description: In each trial, participants are presented with two tones separated by 1200 ms (the standard interval), a 1s delay, then a comparison pair of tones. The time interval of the second tone pair will be either equal to (E-condition), longer than (L-condition), or shorter than (S-condition) that of the first pair. Participants are asked to indicate using a keyboard whether the second time interval is equal, longer, or shorter than the first. The tones for all conditions were 700Hz in frequency, 50ms in duration, and presented binaurally via headphones. Participants completed 15 trials during each pre- or post-TMS session for a total of up to 90 total trials across the three study visits. Prior to each IDT session, participants performed a practice run consisting of six trials. The primary outcome for this task was overall accuracy (proportion of correct responses).
Time Frame: In each of the 3 study visits (separated by at least 36h), participants undergo (a) pre-TMS assessments (15-20min), (b) TMS (15min), and (c) post-TMS assessments (15-20min). Approximately 30-45 min separate the pre- and post-TMS task performances.
Population: Cross-over design in which patients were assigned to 3 sessions of cerebellar TBS: one session each of iTBS, cTBS, and sham TBS. Analyses were conducted for all participants (patients who completed at least one study visit; n=26) as well as for completers only (patients who completed all 3 study visits; n=20; results not reported here). The fields for "overall number of participants analyzed" (above) indicate all participants who completed each of the sessions (iTBS, cTBS, sham TBS).
Measure: Mean (Standard Deviation); unit: accuracy (proportion correct)
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
accuracy (proportion correct)
  Pre-TBS | .503 (.156) | .521 (.183) | .456 (.141)
  Post-TBS | .479 (.128) | .514 (.145) | .525 (.174)
  Change in accuracy (post-pre) | -.024 (.175) | -.006 (.163) | .069 (.198)
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Sham TBS; Conducted a mixed effects analysis, with IDT accuracy as the dependent variable and time (pre, post), condition (iTBS vs. sham, cTBS vs. sham), and the interaction of time x condition (time x iTBS, time x cTBS) as the independent variables. P-value here is for the iTBS (vs. sham) x time interaction; Test type: Equivalence — Tested the null hypothesis of no difference between iTBS and sham TBS on IDT accuracy; p = 0.51, Mixed Models Analysis — Significance threshold of p < 0.05, two-sided; Model included time (pre, post), condition (iTBS vs. sham, cTBS vs. sham), and the interaction of time x condition (time x iTBS, time x cTBS); Beta coefficient for timexiTBS interact = -.099, 95% CI 2-sided [-.1989 to .0002], Standard Error of Mean .051
Statistical Analysis 2: Comparison: Continuous TBS (cTBS) vs Sham TBS; Conducted a mixed effects analysis, with IDT accuracy as the dependent variable and time (pre, post), condition (iTBS vs. sham, cTBS vs. sham), and the interaction of time x condition (time x iTBS, time x cTBS) as the independent variables. P-value here is for the cTBS (vs. sham) x time interaction; Test type: Equivalence — Tested the null hypothesis of no difference between iTBS and sham TBS on IDT accuracy; p = 0.143, Mixed Models Analysis — Significance threshold of p < 0.05, two-sided; [statistical method as in outcome 1, analysis 1]; Beta coefficient for timexcTBS interact = -.0757, 95% CI 2-sided [-.1770 to .0256], Standard Error of Mean .052

2. Primary Outcome: Change (Δ) in Accuracy of N-back Working Memory Task Pre- and Post-TMS
Description: Participants are presented with a series of words or numbers and prompted to indicate as quickly as possible whether the currently presented stimulus is the same as the one presented n-stimuli previously. For example, in a 2-back task a subject would be asked to indicate whether the current stimulus was identical to that presented 2 stimuli before. To increase the likelihood of detecting change in task performance with each TMS condition (and minimize potential ceiling or floor effects), the difficulty level was individualized so that each participant performed at approximately 80% accuracy; during the "pre" session of the first study visit, a trial session established the difficulty level, i.e., how many presentations back (n-stimuli) at which the task would start. After the trial session, a session with 50 presentations was carried out and recorded whether the response was correct (accuracy) and the time from presentation to response (reaction time).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: accuracy (proportion correct)
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
accuracy (proportion correct)
  Pre-TBS | 0.780 (0.0144) | 0.753 (0.0156) | 0.775 (0.0143)
  Post-TBS | 0.795 (0.0138) | 0.778 (0.0147) | 0.784 (0.0139)
  Ratio (post/pre) | 1.10 (.074) | 1.15 (.077) | 1.05 (.065)
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Sham TBS; Conducted a generalized linear mixed model fit by maximum likelihood (Laplace Approximation) ['glmerMod' in R] with binomial (logit) distribution. N-back accuracy was the dependent variable. Time (pre vs. post), condition (iTBS vs. sham, cTBS vs. sham), and the interaction of time x condition (time x iTBS, time x cTBS) were the independent variables. P-value here is for the iTBS (vs. sham) x time interaction; Test type: Equivalence — Tested the null hypothesis of no difference between iTBS and sham TBS on N-back accuracy; p = .626, Mixed Models Analysis — Significance threshold was p < 0.05, two-sided; Beta coefficient for timexiTBS interact = -.0446
Statistical Analysis 2: Comparison: Continuous TBS (cTBS) vs Sham TBS; Conducted a generalized linear mixed model fit by maximum likelihood (Laplace Approximation) ['glmerMod' in R] with binomial (logit) distribution. N-back accuracy was the dependent variable. Time (pre vs. post), condition (iTBS vs. sham, cTBS vs. sham), and the interaction of time x condition (time x iTBS, time x cTBS) were the independent variables. P-value here is for the cTBS (vs. sham) x time interaction; Test type: Equivalence — Tested the null hypothesis of no difference between cTBS and sham TBS on N-back accuracy; p = 0.322, Mixed Models Analysis — Significance threshold was p < 0.05, two-sided; Beta coefficient for timexcTBS interact = -0.0903

3. Primary Outcome: Change (Δ) in Reaction Time (RT) of N-back Working Memory Task Pre- and Post-TMS
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
ms
  Pre-TBS | 831 (13.29) | 862 (14.62) | 901 (11.63)
  Post-TBS | 817 (10.66) | 886 (10.80) | 877 (9.16)
  Change in RT (post-pre) | -14 (8.90) | 24.0 (11.46) | -23.8 (7.41)
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Conducted a generalized linear mixed model fit by maximum likelihood (Laplace Approximation) ['glmerMod' in R] with gamma distribution. N-back reaction time (RT) was the dependent variable. Time (pre vs. post), condition (iTBS vs. sham, cTBS vs. sham), and the interaction of time x condition (time x iTBS, time x cTBS) were the independent variables. P-value here is for the iTBS (vs. sham) x time interaction; Test type: Equivalence — Tested the null hypothesis of no difference between iTBS and sham TBS on N-back accuracy; p = 0.1118, Mixed Models Analysis — Significance threshold of p < 0.05, two-sided; Beta coefficient for timexiTBS interact = -9.797
Statistical Analysis 2: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Conducted a generalized linear mixed model fit by maximum likelihood (Laplace Approximation) ['glmerMod' in R] with gamma distribution. N-back reaction time (RT) was the dependent variable. Time (pre vs. post), condition (iTBS vs. sham, cTBS vs. sham), and the interaction of time x condition (time x iTBS, time x cTBS) were the independent variables. P-value here is for the cTBS (vs. sham) x time interaction; Test type: Equivalence — Tested the null hypothesis of no difference between cTBS and sham TBS on N-back accuracy; p = 0.00000009, Mixed Models Analysis — Significance threshold was p < 0.05, two-sided; Beta coefficient for timexcTBS interact = -47.764

4. Primary Outcome: Change (Δ) in Symptoms (Depressed Mood)
Description: Participants will take a brief computerized survey pre- and post-TMS, in which they will be presented with visual analogue scales (VAS, range 0-100, 0=absent, 100=most severe) and asked to indicate current levels of depression, anxiety, euphoria, auditory hallucinations, visual hallucinations, paranoia, referential thinking, and delusions of control. The VAS format will allow participants to self-report ratings quickly and easily with simple mouse clicks.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
score on a scale
  Pre-TBS | 22.5 [0 to 70] | 37 [0 to 91] | 16 [0 to 70]
  Post-TBS | 19.5 [0 to 72] | 42 [0 to 71] | 4 [0 to 76]
  Change in VAS score (post-pre) | 0 [-31 to 63] | 0 [-41 to 26] | 0 [-43 to 7]
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Test type: Equivalence — Tested the null hypothesis that there is no effect of condition (iTBS, cTBS, sham) on pre-post change in VAS scores; p = 0.910, Friedman test — Given the exploratory nature of this pilot study, we set the significance threshold at p < 0.05, two-sided, without correcting for eight comparisons; Non-parametric repeated measures ANOVA
Statistical Analysis 2: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; We explored the association between interval discrimination task (IDT) performance (accuracy) and each symptom self-rating (here, depressed mood). We conducted a mixed effects regression analysis to test the null hypothesis of no association. Model included time (pre, post) and condition (iTBS vs. sham, cTBS vs. sham) in addition to symptom rating as independent variables, and IDT performance accuracy as the dependent variable; Test type: Other — Given the exploratory nature of this pilot study, we set the significance threshold at p <0.05, two-sided, without correcting for eight comparisons; p = 0.243, Mixed Models Analysis; beta coefficient for depressed mood = 0.00071, 95% CI 2-sided [-0.00048 to 0.00190]

5. Primary Outcome: Change (Δ) in Symptoms (Anxiety)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
score on a scale
  Pre-TBS | 22 [0 to 73] | 50 [0 to 87] | 23 [0 to 74]
  Post-TBS | 4 [0 to 75] | 30 [0 to 77] | 5 [0 to 73]
  Change in VAS score (post-pre) | -2.5 [-50 to 24] | -1 [-40 to 32] | 0 [-30 to 22]
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Test type: Equivalence — Tested the null hypothesis that there is no effect of condition (iTBS, cTBS, sham) on pre-post change in VAS scores; p = 0.830, Friedman test — [p-value comment as in outcome 4, analysis 1]; Non-parametric repeated measures ANOVA
Statistical Analysis 2: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; We explored the association between interval discrimination task (IDT) performance (accuracy) and each symptom self-rating (here, anxiety). We conducted a mixed effects regression analysis to test the null hypothesis of no association. Model included time (pre, post) and condition (iTBS vs. sham, cTBS vs. sham) in addition to symptom rating as independent variables, and IDT performance accuracy as the dependent variable; Test type: Other; p = 0.284, Mixed Models Analysis — Given the exploratory nature of this pilot study, we set the significance threshold at p <0.05, two-sided, without correcting for eight comparisons; beta coefficient for anxiety = -0.00063, 95% CI 2-sided [-0.00179 to 0.00052]

6. Primary Outcome: Change (Δ) in Symptoms (Elated Mood)
Description: Participants will take a brief computerized survey pre- and post-TMS, in which they will be presented with visual analogue scales (VAS, range 0-100, 0=absent/no elation, 100=most severe) and asked to indicate current levels of depression, anxiety, euphoria, auditory hallucinations, visual hallucinations, paranoia, referential thinking, and delusions of control. Higher VAS scores for elation indicate more elation (suggestive of mania). The VAS format will allow participants to self-report ratings quickly and easily with simple mouse clicks.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
score on a scale
  Pre-TBS | 6 [0 to 54] | 2 [0 to 51] | 1 [0 to 53]
  Post-TBS | 8.5 [0 to 60] | 0 [0 to 57] | 1 [0 to 40]
  Change in VAS score (post-pre) | 0 [-54 to 49] | 0 [-24 to 51] | 0 [-50 to 37]
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Test type: Equivalence — Tested the null hypothesis that there is no effect of condition (iTBS, cTBS, sham) on pre-post change in VAS scores; p = 0.755, Friedman test — [p-value comment as in outcome 4, analysis 1]; Non-parametric repeated measures ANOVA
Statistical Analysis 2: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; We explored the association between interval discrimination task (IDT) performance (accuracy) and each symptom self-rating (here, elated mood). We conducted a mixed effects regression analysis to test the null hypothesis of no association. Model included time (pre, post) and condition (iTBS vs. sham, cTBS vs. sham) in addition to symptom rating as independent variables, and IDT performance accuracy as the dependent variable; Test type: Other; p = 0.317, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; beta coefficient for elated mood = -0.00070, 95% CI 2-sided [-0.00208 to 0.00067]

7. Primary Outcome: Change (Δ) in Symptoms (Auditory Hallucinations)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
score on a scale
  Pre-TBS | 0 [0 to 65] | 0 [0 to 50] | 0 [0 to 70]
  Post-TBS | 0 [0 to 49] | 0 [0 to 50] | 0 [0 to 65]
  Change in VAS score (post-pre) | 0 [-44 to 1] | 0 [-9 to 48] | 0 [-9 to 50]
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Test type: Equivalence — Tested the null hypothesis that there is no effect of condition (iTBS, cTBS, sham) on pre-post change in VAS scores; p = .035, Friedman test — [p-value comment as in outcome 4, analysis 1]; Non-parametric repeated measures ANOVA
Statistical Analysis 2: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; We explored the association between interval discrimination task (IDT) performance (accuracy) and each symptom self-rating (here, auditory hallucinations). We conducted a mixed effects regression analysis to test the null hypothesis of no association. Model included time (pre, post) and condition (iTBS vs. sham, cTBS vs. sham) in addition to symptom rating as independent variables, and IDT performance accuracy as the dependent variable; Test type: Other; p = 0.028, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; beta coefficient for auditory hallucinat = 0.00195, 95% CI 2-sided [0.00021 to 0.00369]

8. Primary Outcome: Change (Δ) in Symptoms (Visual Hallucinations)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
score on a scale
  Pre-TBS | 0 [0 to 52] | 0 [0 to 79] | 0 [0 to 50]
  Post-TBS | 0 [0 to 53] | 0 [0 to 56] | 0 [0 to 50]
  Change in VAS score (post-pre) | 0 [-22 to 9] | 0 [-29 to 8] | 0 [-13 to 50]
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Test type: Equivalence — Tested the null hypothesis that there is no effect of condition (iTBS, cTBS, sham) on pre-post change in VAS scores; p = .748, Friedman test — [p-value comment as in outcome 4, analysis 1]; Non-parametric repeated measures ANOVA
Statistical Analysis 2: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; We explored the association between interval discrimination task (IDT) performance (accuracy) and each symptom self-rating (here, visual hallucinations). We conducted a mixed effects regression analysis to test the null hypothesis of no association. Model included time (pre, post) and condition (iTBS vs. sham, cTBS vs. sham) in addition to symptom rating as independent variables, and IDT performance accuracy as the dependent variable; Test type: Other; p = 0.685, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; beta coefficient for visual hallucinatio = -0.00039, 95% CI 2-sided [-0.00230 to 0.00151]

9. Primary Outcome: Change (Δ) in Symptoms (Paranoid Ideation)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
score on a scale
  Pre-TBS | 0 [0 to 55] | 0 [0 to 63] | 0 [0 to 71]
  Post-TBS | 0 [0 to 50] | 0 [0 to 59] | 0 [0 to 100]
  Change in VAS score (post-pre) | 0 [-24 to 41] | 0 [-43 to 3] | 0 [-18 to 43]
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Test type: Equivalence — Tested the null hypothesis that there is no effect of condition (iTBS, cTBS, sham) on pre-post change in VAS scores; p = .020, Friedman test — [p-value comment as in outcome 4, analysis 1]; Non-parametric repeated measures ANOVA
Statistical Analysis 2: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; We explored the association between interval discrimination task (IDT) performance (accuracy) and each symptom self-rating (here, paranoid ideation). We conducted a mixed effects regression analysis to test the null hypothesis of no association. Model included time (pre, post) and condition (iTBS vs. sham, cTBS vs. sham) in addition to symptom rating as independent variables, and IDT performance accuracy as the dependent variable; Test type: Other; p = 0.597, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; beta coefficient for paranoid ideation = 0.00040, 95% CI 2-sided [-0.00108 to 0.00188]

10. Primary Outcome: Change (Δ) in Symptoms (Ideas/Delusions of Reference)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
score on a scale
  Pre-TBS | 0 [0 to 55] | 0 [0 to 51] | 0 [0 to 53]
  Post-TBS | 0 [0 to 50] | 0 [0 to 54] | 0 [0 to 53]
  Change in VAS score (post-pre) | 0 [-5 to 22] | 0 [-50 to 3] | 0 [0 to 11]
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Test type: Equivalence — Tested the null hypothesis that there is no effect of condition (iTBS, cTBS, sham) on pre-post change in VAS scores; p = .237, Friedman test — [p-value comment as in outcome 4, analysis 1]; Non-parametric repeated measures ANOVA
Statistical Analysis 2: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; We explored the association between interval discrimination task (IDT) performance (accuracy) and each symptom self-rating (here, ideas/delusions of reference). We conducted a mixed effects regression analysis to test the null hypothesis of no association. Model included time (pre, post) and condition (iTBS vs. sham, cTBS vs. sham) in addition to symptom rating as independent variables, and IDT performance accuracy as the dependent variable; Test type: Other; p = 0.178, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; beta coefficient for ideas/del of refere = -0.00142, 95% CI 2-sided [-0.00350 to 0.00065]

11. Primary Outcome: Change (Δ) in Symptoms (Delusions of Control)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
Number analyzed (Participants) | 22 | 21 | 25
score on a scale
  Pre-TBS | 0 [0 to 50] | 0 [0 to 25] | 0 [0 to 3]
  Post-TBS | 0 [0 to 29] | 0 [0 to 73] | 0 [0 to 11]
  Change in VAS score (post-pre) | 0 [-48 to 28] | 0 [-24 to 48] | 0 [-2 to 11]
Statistical Analysis 1: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; Test type: Equivalence — Tested the null hypothesis that there is no effect of condition (iTBS, cTBS, sham) on pre-post change in VAS scores; p = .330, Friedman test — [p-value comment as in outcome 4, analysis 1]; Non-parametric repeated measures ANOVA
Statistical Analysis 2: Comparison: Intermittent TBS (iTBS) vs Continuous TBS (cTBS) vs Sham TBS; We explored the association between interval discrimination task (IDT) performance (accuracy) and each symptom self-rating (here, delusions of control). We conducted a mixed effects regression analysis to test the null hypothesis of no association. Model included time (pre, post) and condition (iTBS vs. sham, cTBS vs. sham) in addition to symptom rating as independent variables, and IDT performance accuracy as the dependent variable; Test type: Other; p = 0.777, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; beta coefficient for delusions of contro = -0.00038, 95% CI 2-sided [-0.00305 to 0.00228]

ADVERSE EVENTS:
Time Frame: Varied. Approximately one-month time frame (mean 11.6 ± 6.6, range 4-28 days). Participants were monitored for adverse events from enrollment to end of study participation.
Arm/Group | Intermittent TBS (iTBS) | Continuous TBS (cTBS) | Sham TBS
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/25
Other Adverse Events (participants affected / at risk) | 2/22 | 0/21 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent TBS (iTBS) (N=22) | Continuous TBS (cTBS) (N=21) | Sham TBS (N=25)
Discomfort from TMS (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
(1) Small sample size. (2) Statistical analyses uncorrected for multiple comparisons. (3) Sample consisted mostly of stable outpatients with low symptom severity. (4) IDT task difficulty was not adjusted to participant performance. (5) Negative symptoms were not evaluated. However, acute changes in negative symptoms (which tend to be trait-like phenomena) are more challenging to measure. (6) Study did not include any biological markers (e.g., imaging) by which to measure TBS effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT02642029/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT02642029/SAP_001.pdf